CLINICAL TRIAL: NCT05840367
Title: Mothers' Experience of Category 1 Cesarean Section - in a Hospital Where the Partner is Present in the Operating Room. A Qualitative Study.
Brief Title: Mothers' Experience of Category 1 Cesarean Section
Status: Recruiting | Type: Observational
Sponsor: Sygehus Lillebaelt (Other)
Collaborators: University of Southern Denmark, Department of Regional Health Research (Unknown)
Responsible Party: Principal Investigator, Helene Korvenius Nedergaard, MD, PhD, Sygehus Lillebaelt
Other Study IDs: 972294863
Record Dates: First submitted 2023-04-18; First posted 2023-05-03 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Partner present in the operation room — The partner (father, co-mother or other close relative present for the birth) is present in the operation room during the entire category 1 cesarean section. This is standard clinical practice in this particular hospital since June 2021.

SUMMARY:
The aim of this qualitative prospective study is to investigate how mothers experience a category 1 cesarean section in a hospital where the partner is present in the operation room during the entire process (induction of general anestesia, cesarean section, possible resuscitation of newborn).

Mothers will be included in the study, if they wish to participate, on day 1 or 2 following the cesarean section and a brief, structured interview will be held concerning her experience of the cesarean section.

Clinical baseline data regarding the mother, the cesarean section and the infant will be collected from patients files.

Mothers will be contacted again three months after the cesarean section, and a semi-structured interview will be held via telephone. At the end of the interview a screening for posttraumatic stress will be performed, using the PTSD-8 tool. The interviews will be recorded and transscribed verbatim.

Content of interviews will be analysed using manifest content analysis. NVivo software will be used for coding interviews.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who had a category 1 cesarean section in Kolding Hospital, Denmark during a 1-year period

Exclusion Criteria:

* Not speaking/understanding Danish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to include all mothers who undergoes a category 1 cesarean section in Kolding Hospital, Denmark, during a 1-year period. Mothers will be approached for inclusion in the study regardless of the outcome of the infant.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mothers' experience of the category 1 cesarean section | Three months after the cesarean section
  Qualitative analysis of data regarding mothers' experience of a category 1 cesarean section in a hospital where the partner is present in the operation room.
  Semi-structured interviews will be held, recorded digitally and transscribed. Content will be analysed qualitatively using manifest content analysis, and major themes as well as sub-themes will be identified, describing mothers' experience with the category 1 cesarean section.

SECONDARY OUTCOMES:
PTSD | Three months after the cesarean section
  Occurence of posttraumatic stress as evaluated using the PTSD-8 tool (in Danish)

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Brøchner, MD, Associate Professor, Study Chair — Lillebaelt Hospital Kolding, Department of Anesthesiology and Intensive Care, and University of Southern Denmark, Department of Regional Health Research
Locations (1):
- Lillebaelt Hospital, Kolding, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared.